CLINICAL TRIAL: NCT06534892
Title: A Phase 3b, Randomized, Open Label, Multicountry, Multi-center, Extension and Crossover Vaccination Study to Evaluate the Immunogenicity and Safety of Different Revaccination Schedules and Persistence of a Single Dose of the RSVPreF3 OA Vaccine in Adults Aged 60 Years and Above Who Participated in the RSV OA=ADJ-006 Study
Brief Title: An Extension and Crossover Vaccination Study on the Immune Response and Safety of a Vaccine Against Respiratory Syncytial Virus Given to Adults 60 Years of Age and Above Who Participated in RSV OA=ADJ-006 Study
Acronym: RSV OA=ADJ=012
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 222090; 2023-509762-38-00 (Other: EU CTR Number)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus (RSV); Older adults; RSVPreF3 OA vaccine; Immunogenicity; Safety; RSV Season
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: This is an extension and crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RSV_PreS4 (Experimental): Participants in this group will receive 1 dose of RSVPreF3 OA vaccine before RSV Season 4.
  Interventions: Biological: RSVPreF3 OA vaccine
- RSV_PreS5 (Experimental): Participants in this group will receive 1 dose of RSVPreF3 OA vaccine before RSV Season 5.
  Interventions: Biological: RSVPreF3 OA vaccine
- RSV_1Dose (No Intervention): Participants in this group will not receive any additional dose of RSV PreF3 OA vaccine.
- Crossover (Experimental): Participants in this group will receive a single dose of RSVPreF3 OA vaccine.
  Interventions: Biological: RSVPreF3 OA vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA vaccine — RSVPreF3 OA vaccine administered at different timepoints (revaccination groups) or for the first time (crossover group)
  Arms: Crossover; RSV_PreS4; RSV_PreS5

SUMMARY:
The purpose of this study is:

* To investigate the optimal timing for revaccination after the initial RSVPreF3 OA vaccine dose,
* To evaluate the long-term immune persistence and safety up to 5 consecutive RSV seasons (approximately 60 months) of a single dose of RSVPreF3 OA vaccine,
* To give the opportunity to participants who received only placebo in the RSVOA=ADJ- 006 study, to receive a dose of the RSVPreF3 OA vaccine and collect additional safety information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who were previously enrolled in the RSV OA=ADJ-006 study and received placebo (Placebo group) or a single dose of the RSVPreF3 OA vaccine (RSV_1dose group).
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, attend regular phone calls/study site visits, ability to access and utilize a phone or other electronic communications).
* Written or witnessed informed consent obtained from the participant prior to performance of any study specific procedure.
* Participants who are medically stable in the opinion of the investigator at study entry. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study.

Exclusion Criteria:

Medical Conditions:

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Hypersensitivity to latex.
* Serious or unstable chronic illness.
* Recurrent or un-controlled neurological disorders or seizures.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any other medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Any history of dementia or any medical condition that moderately or severely impairs cognition and understanding of the informed consent form and/or study procedures.
* Participants who experienced an SAE or pIMD from first study intervention administration in the RSV OA=ADJ-006 study until enrollment in this study that was considered to be possibly or probably related to the study vaccine or non-study concomitant vaccines, either by the investigator or the sponsor, including hypersensitivity reactions.
* Participants with a new onset of a pIMD or exacerbation of a pIMD from first study intervention administration in the RSV OA=ADJ-006 study until enrollment in this study, that, in the opinion of the investigator, exposes the participant to unacceptable risk from subsequent vaccination.

Prior/Concomitant Therapy:

• Use of any investigational or non-registered product other than the study vaccine during the period beginning 30 days before the first dose of study vaccine, or planned use during the study period. • Previous vaccination with an RSV vaccine (investigational or licensed vaccine) and/or planned administration of an RSV vaccine during the study period other than the RSVPreF3 OA vaccine administered during the RSV OA=ADJ-006 study.

Prior/Concurrent Clinical Study Experience:

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.

Other Exclusion Criteria:

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Participation of any study personnel or their immediate dependents, family, or household members.
* Bedridden participants.

Specific exclusion criteria for Crossover group:

• Planned or administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after study intervention administration, with the exception of COVID vaccines which can be administered up to 14 days before or from 14 days after study vaccination. Inactivated seasonal influenza vaccines can be co-administered or administered at any time.

Specific exclusion criteria for RSV_PreS4, RSV_PreS5 and RSV_1Dose groups:

* Planned or administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after study intervention administration, with the exception of COVID vaccines and inactivated seasonal influenza vaccines which can be administered up to 14 days before or from 14 days after study intervention administration.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the first study visit or planned administration during the study period.
* Chronic administration of immunosuppressants or other immunemodifying drugs during the period starting 90 days prior to the first study visit or planned administration during the study period. For corticosteroids, this will mean prednisone >= 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10212 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
RSV-A neutralizing titers expressed as Geometric mean titers (GMTs) in RSV_PreS4 group at Day 1 | At Day 1
RSV-A neutralizing titers expressed as GMTs in RSV_PreS4 group at Day 31 | At Day 31
RSV-B neutralizing titers expressed as GMTs in RSV_PreS4 group at Day 1 | At Day 1
RSV-B neutralizing titers expressed as GMTs in RSV_PreS4 group at Day 31 | At Day 31
RSV-A neutralizing titers expressed as Mean geometric increase (MGI) in RSV_PreS4 group | From Day 1 to Day 31
RSV-B neutralizing titers expressed as MGI in RSV_PreS4 group | From Day 1 to Day 31
Percentage of participants with RSV-A neutralizing titers greater than or equal to (>=) cut-off in RSV_PreS4 group at Day 1 | At Day 1
Percentage of participants with RSV-A neutralizing titers >= cut-off in RSV_PreS4 group at Day 31 | At Day 31
Percentage of participants with RSV-B neutralizing titers >=cut-off in RSV_PreS4 group at Day 1 | At Day 1
Percentage of participants with RSV-B neutralizing titers >=cut-off in RSV_PreS4 group at Day 31 | At Day 31
Percentage of participants with seroresponse rate (SRR) for RSV-A neutralizing titers in RSV_PreS4 group | At Day 31
Percentage of participants with SRR for RSV-B neutralizing titers in RSV_PreS4 group | At Day 31
RSV-A neutralizing titers expressed as GMT in RSV_PreS5 group at Day 1 | At Day 1
RSV-A neutralizing titers expressed as GMT in RSV_PreS5 group at Month 12 | At Month 12
RSV-A neutralizing titers expressed as GMT in RSV_PreS5 group at Month 13 | At Month 13
RSV-A neutralizing titers expressed as GMT in RSV_PreS5 group at Month 24 | At Month 24
RSV-B neutralizing titers expressed as GMTs in RSV_PreS5 group at Day 1 | At Day 1
RSV-B neutralizing titers expressed as GMTs in RSV_PreS5 group at Month 12 | At Month 12
RSV-B neutralizing titers expressed as GMTs in RSV_PreS5 group at Month 13 | At Month 13
RSV-B neutralizing titers expressed as GMTs in RSV_PreS5 group at Month 24 | At Month 24
RSV-A neutralizing titers expressed as MGI in RSV_PreS5 group from Month 12 to Month 13 | From Month 12 to Month 13
RSV-A neutralizing titers expressed as MGI in RSV_PreS5 group from Month 12 to Month 24 | From Month 12 to Month 24
RSV-B neutralizing titers expressed as MGI in RSV_PreS5 group from Month 12 to Month 13 | From Month 12 to Month 13
RSV-B neutralizing titers expressed as MGI in RSV_PreS5 group from Month 12 to Month 24 | From Month 12 to Month 24
Percentage of participants with RSV-A neutralizing titers >=cut-off in RSV_PreS5 group at Day 1 | At Day 1
Percentage of participants with RSV-A neutralizing titers >=cut-off in RSV_PreS5 group at Month 12 | At Month 12
Percentage of participants with RSV-A neutralizing titers >=cut-off in RSV_PreS5 group at Month 13 | At Month 13
Percentage of participants with RSV-A neutralizing titers >=cut-off in RSV_PreS5 group at Month 24 | At Month 24
Percentage of participants with RSV-B neutralizing titers >=cut-off in RSV_PreS5 group at Day 1 | At Day 1
Percentage of participants with RSV-B neutralizing titers >=cut-off in RSV_PreS5 group at Month 12 | At Month 12
Percentage of participants with RSV-B neutralizing titers >=cut-off in RSV_PreS5 group at Month 13 | At Month 13
Percentage of participants with RSV-B neutralizing titers >=cut-off in RSV_PreS5 group at Month 24 | At Month 24
Percentage of participants with seroresponse rate (SRR) for RSV-A neutralizing titers in RSV_PreS5 group | At Month 13
Percentage of participants with SRR for RSV-B neutralizing titers in RSV_PreS5 group | At Month 13

SECONDARY OUTCOMES:
RSV-A neutralizing titers expressed as GMTs in RSV_1Dose group | At Day 1, Month 12 and at Month 24
RSV-B neutralizing titers expressed as GMTs in RSV_1Dose group | At Day 1, Month 12 and at Month 24
Percentage of participants with RSV-A neutralizing titers >= cut-off in RSV_1Dose group | At Day 1, Month 12 and at Month 24
Percentage of participants with RSV-B neutralizing titers >= cut-off in RSV_1Dose group | At Day 1, Month 12 and at Month 24
Number of participants with unsolicited adverse events | At Day 30 post vaccination
Number of participants with any serious adverse events (SAEs) | From day of vaccination and up to 6 months post each vaccine administration
Number of participants with SAEs related to study intervention | From Day 1 and up to end of study
Number of participants with any potential immune-mediated disease (pIMDs) | From day of vaccination and up to 6 months post each vaccine administration
Number of participants with pIMDs related to study intervention | From Day 1 and up to end of study
Number of participants with fatal SAEs | From Day 1 and up to end of study

CONTACTS AND LOCATIONS:
Locations (213):
- United States (53):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lake City, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, The Villages, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Mishawaka, Indiana
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Richfield, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Keller, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Norfolk, Virginia
- Australia (8):
  - GSK Investigational Site, Botany, New South Wales
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Taringa, Queensland
  - GSK Investigational Site, Tarragindi, Queensland
  - GSK Investigational Site, Camberwell, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Spearwood, Western Australia
- Belgium (10):
  - GSK Investigational Site, Diepenbeek
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Erpent
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Ieper
  - GSK Investigational Site, Kluisbergen
  - GSK Investigational Site, Linkebeek
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Tremelo
- Canada (19):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London-Ontario, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Estonia (3):
  - GSK Investigational Site, Paide
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (8):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Germany (22):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dachau
  - GSK Investigational Site, Dippoldiswalde
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Freital
  - GSK Investigational Site, Goch
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Hochheim am Main
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Schenefeld
  - GSK Investigational Site, Wallerfing
  - GSK Investigational Site, Wangen
  - GSK Investigational Site, Witten
  - GSK Investigational Site, Würzburg
- Italy (11):
  - GSK Investigational Site, Alessandria
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Belluno
  - GSK Investigational Site, Ferrara
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Negrar Verona
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pessione - Chieri to
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Siena
- Japan (9):
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamagata
  - GSK Investigational Site, Yamaguchi
- Mexico (9):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, León
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, Oaxaca City
  - GSK Investigational Site, Querétaro
  - GSK Investigational Site, RM Pharmamexico CITY
  - GSK Investigational Site, San Luis Potosí City
- New Zealand (6):
  - GSK Investigational Site, Grafton Auckland
  - GSK Investigational Site, Hawke's Bay
  - GSK Investigational Site, Kapiti
  - GSK Investigational Site, Palmerston North
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Wellington
- Poland (10):
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (7):
  - GSK Investigational Site, Gatchina, Leningradskaya Oblast'
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, StPetersburg
  - GSK Investigational Site, Yekaterinburg
- South Africa (7):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Moloto South
  - GSK Investigational Site, Reiger Park
  - GSK Investigational Site, Tembisa
- South Korea (8):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si Kyunggi-do 14584
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Gyeonggi-do
- Spain (5):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- United Kingdom (18):
  - GSK Investigational Site, Bebington
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bradford on Avon Wiltsh
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Corby
  - GSK Investigational Site, Eynsham
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hexham
  - GSK Investigational Site, Lancashire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Orpington
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Peterborough
  - GSK Investigational Site, Royal Leamington Spa
  - GSK Investigational Site, Thetford
  - GSK Investigational Site, Witney

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.